CLINICAL TRIAL: NCT00392470
Title: Neoadjuvant Conformal Radiotherapy and Concomitant CPT-11 and EGFR Inhibition With Cetuximab in Patients With Rectal Cancer Phase I Study
Brief Title: Radiation Therapy, Irinotecan, and Cetuximab in Treating Patients Who Are Undergoing Surgery for Stage III or Stage IV Rectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000512816; CHUV-CEPO-CORCC-204-5; EU-20645; PFIZER-CHUV-CAPO-CARK-204-5; MERCK-CHUV-CAPO-CARK-204-5
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2008-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Irinotecan; Neoadjuvant Therapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Biological: cetuximab
Drug: irinotecan hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: 3-dimensional conformal radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving radiation therapy together with irinotecan and cetuximab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan when given together with cetuximab and radiation therapy in treating patients who are undergoing surgery for stage III or stage IV rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of irinotecan hydrochloride and cetuximab in patients with stage III or IV rectal cancer undergoing conformal or intensity-modulated radiotherapy.

Secondary

* Determine the rate of pathologic response and histological degree of tumor regression in patients treated with this regimen.
* Determine the complete resection rate (R0) in patients treated with this regimen.
* Determine the sphincter preservation rate in patients treated with this regimen.
* Determine the 30-day postoperative complication rate in patients treated with this regimen.
* Determine the local and distant relapse rate and site of disease failure in patients treated with this regimen.
* Estimate the predictive value of fludeoxyglucose F 18 positron emission tomography/CT scan for treatment response compared to endoscopic ultrasonography (EUS), CT scan, and MRI in patients treated with this regimen.
* Determine the late toxicity of this regimen in these patients.
* Determine the clinical (radiological) tumor response (i.e., MRI, CT scan, EUS) in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of irinotecan hydrochloride.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, and 43 followed by irinotecan hydrochloride IV over 30 minutes on days 1, 8, 15, 22, and 29. Patients also undergo conformal radiotherapy or intensity-modulated radiotherapy on days 1-5 for 5 weeks. Patients undergo radical surgery 3-4 weeks after completion of neoadjuvant therapy.

Cohorts of 3-6 patients receive escalating doses of irinotecan hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * T3-4 and/or N+ (stage IIIB, IIIC, or IV disease)
* Liver or lung metastasis allowed
* No recurrent disease

PATIENT CHARACTERISTICS:

* WHO performance status 0 or 1
* Hematologic, liver, and renal function normal
* Considered fit for chemotherapy, radiotherapy, and surgery
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No symptomatic heart disease or myocardial infarction during the past 6 months
* No chronic inflammatory bowel disease
* No malignant tumor during the past 5 years except for completely surgically resected carcinoma of the cervix or squamous cell carcinoma of the skin
* No other concurrent malignant tumor

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for rectal cancer
* No prior radiotherapy to the pelvis

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Radiological (clinical) tumor response before surgery
Pathologic response rate and histological degree of tumor regression as measured by Mandard TRG score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Montemurro, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (3):
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Institut Ludwig de Recherche sur le Cancer, Épalinges
  - Centre Hospitalier Universitaire Vaudois, Lausanne